CLINICAL TRIAL: NCT02399124
Title: ICE-SECRET PROSENSE™ Cryotherapy For Renal Cell Carcinoma Trial
Brief Title: Post Marketing Surveillance for PROSENSE™ a Cryotherapy Treatment of Renal Cell Carcinoma
Acronym: ICE-SECRET
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IceCure Medical Ltd. (Industry)
Collaborators: Bnai Zion Medical Center (Other Government); Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICMRC-01
Record Dates: First submitted 2015-01-27; First posted 2015-03-26 (Estimated); Last update posted 2026-01-06 (Actual); Status verified 2025-04

CONDITIONS: Renal Cell Carcinoma
Keywords: RCC; Renal Cell Carcinoma; Kidney tumors
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single arm, open label, treatment (Other): single arm, open label, treatment; ProSenseTM Cryoablation treatment, post marketing surveillance
  Interventions: Device: PROSENSE™

INTERVENTIONS:
Device: PROSENSE™ — single arm, open label, PROSENSE™ treatment

SUMMARY:
This experiment is designed for post marketing data collection of a cryosurgical system [PROSENSE™ of IceCure Medical], for the treatment of renal cell carcinoma (RCC).

DETAILED DESCRIPTION:
A post marketing data collection of a cryosurgical system [PROSENSE™] of IceCure Medical], for the treatment of renal cell carcinoma (RCC).

ELIGIBILITY:
Inclusion Criteria:

1. Patient is above 18 years old.
2. The patient has enhanced solid mass of renal origin located in the kidney or elsewhere proved by imaging.
3. Patient's mass size is up to 5 cm at its largest dimension.
4. Patient is able to visit the clinic as needed during the 60-month follow-up period following the cryoablation procedure.
5. The patient has been informed of the study and agrees to its provisions, and has signed an IRB approved written informed consent, including data privacy authorization.

Exclusion Criteria:

1. Patients with permanent coagulation disorders or severe medical instability or active infection.
2. Patients with any terminal illness.
3. Patient participating in other trials using drugs or devices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-07 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Success in creating an ice ball that engulfs the whole tumor with 5 mm margins using the ProSense™ as seen under laparoscopic, US or CT imaging during the procedure. | During intervention
  % of procedures with sufficient engulfment
Recurrence free survival | up to 5 years
  % of local recurrence events

SECONDARY OUTCOMES:
Success in verification of the ProSense™ safety as demonstrated by having no complications related to the cryoablation procedure other than the well-known ones. | a follow up visit at 6 weeks, 6 months, 12 months and every 1 year afterwards up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Halachmi Sarel, Prof., Principal Investigator — Bnei Zion Medical Center, Israel
Locations (2):
- Israel (2):
  - Bnei Zion Medical Center, Haifa
  - Shamir Medical Center, Ẕerifin